CLINICAL TRIAL: NCT04685642
Title: Anti-inflmmation Treatment in Mood Disorder and Deep Learning Prediction Model
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 109-2314-B-010 -050 -MY3
Record Dates: First submitted 2020-12-06; First posted 2020-12-28 (Actual); Last update posted 2020-12-28 (Actual); Status verified 2020-12

CONDITIONS: Mood Disorder
Keywords: Anti-inflammatory treatment; depression; bipolar disorder; telomere length; brain imaging
MeSH Terms: conditions — Mood Disorders; Depression; Bipolar Disorder | interventions — Aspirin; Atorvastatin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- non-drug (No Intervention)
- Aspirin (Active Comparator)
  Interventions: Drug: Aspirin
- Statin (Active Comparator)
  Interventions: Drug: Atorvastatin

INTERVENTIONS:
Drug: Aspirin — Aspirin (100mg/day)
  Arms: Aspirin
Drug: Atorvastatin — Atorvastatin (20mg/day)
  Arms: Statin

SUMMARY:
This three-year study will enroll 180 patients with mood disorders (90 patients with major depressive disorder and 90 patients with bipolar disorder) and high pro-inflammatory cytokine levels. They will be randomly assigned to three groups of aspirin, statin and control groups for 12 weeks according to the disease group. The first aim of the study is to compare the efficacy of aspirin and statin in mood disorders. The second aim is to establish a gene-immuno-brain imaging treatment prediction model by deep learning technology, using pretreatment cytokines, neurocognitive function, brain structural/functional connectivity, and telomere length as the predictors.

DETAILED DESCRIPTION:
Multiple lines of evidence support the pathogenic role of neuro-inflammation in mood disorders. Our team has published a series of papers showing the inflammatory cytokines are related to severity of depressive symptoms, could be biomarkers of clinical outcomes, subtype and mood phase of bipolar disorder. Compared with depressive disorder, bipolar disorder is with more severe inflammatory dysregulation, which correlated to brain structure and functional connectivity abnormality. Treatment non-responders tended to have higher baseline inflammatory markers, suggesting that increased levels of inflammation are contributory to treatment resistance. The clinical studies showed that anti-inflammatory drugs combined with traditional treatments, can improve clinical outcomes, including N-Acetylcysteine, infliximab, pioglitazone, celecoxib, aspirin, omega-3 polyunsaturated fatty acids, minocyclin, statin, aspirin. Among them, aspirin and statin have been used for treatment and prevention of cardiovascular metabolic disorders, which are associated with inflammation dysregulation. The clinical and meta-analysis studies of aspirin and statin have shown significant efficacy and good safety. Therefore, aspirin and statin have better clinical feasibility and rationality for augmentation treatment in mood disorders. However, previous anti-inflammatory research is mostly for individual drug studies, comparative research is still quite lacking. In addition, many studies have suggested anti-inflammatory agents will likely be most useful for the subpopulation of patients whose immune dysfunction is a driving pathogenic factor.

In this study, we will establish a prediction model of anti-inflammatory drugs for mood disorder. Recent advances in deep learning have demonstrated its power to learn and recognize complex nonlinear hierarchical patterns based on largescale empirical data. A deep learning algorithm for classification applications such as medical treatment in personalized medicine is a procedure for choosing the best hypothesis from a set of alternatives that fit a set of observations. Our series of studies have shown that the severity of inflammation related with brain structure and functional connectivity abnormalities; which may be the outcome predictors. Another possible predictor may be the chromosome telomere length. Telomeres are located at the end of chromosomes and maintain normal function of chromosomes. Previous studies have found that short telomere length is associated with mood disorder, as well as the inflammatory dysregulation. Therefore, telomere length may be a predictor of anti-inflammatory treatment. The study will be the first comparative study of anti-inflammatory treatment, and establish gene-immuno-brain imaging individualized treatment prediction model. The results will provide important scientific and clinical empirical data for the inflammatory pathophysiology and treatment of mood disorders.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 20 to 65 years old.
2. The baseline pro-inflammatory cytokines level: soluble IL6 receptor (sIL-6)>35,000pg/ml, or CRP>1,500ng/ml, or sTNF-R1>1,000pg/ml.
3. Maintain psychiatric medication for more than three months.
4. Voluntary patients and controls with signed informed consent proved by institutional review board (IRB).

Exclusion Criteria:

1. Patients have used aspirin, statin previously .
2. Patients have gastrointestinal disease, history of gastrointestinal bleeding, hematology coagulation disease, sever liver and renal disease.
3. Patients with schizophrenia, organic brain diseases, mental retardation.
4. Patients with symptoms of substance abuse/dependence (except nicotine dependence) within 3 months.
5. Patients with autoimmune, acute infection and critical medical illnesses .
6. Patients who cannot cooperate the study protocol.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2020-08-24 (Actual); Primary Completion 2023-07-31 (Estimated); Study Completion 2023-07-31 (Estimated)

PRIMARY OUTCOMES:
Reduction rate the clinical symptoms after original treatment combined aspirin or atorvastatin. | baseline, week 4, week 8, week 12
  Treatment Efficacy

SECONDARY OUTCOMES:
The T1-weight | Once on baseline.
  The T1-weight will be taken on a 3T MR scanner (Discovery 750, GE).
The resting fMRI | Once on baseline.
  The resting fMRI will be taken on a 3T MR scanner (Discovery 750, GE).

CONTACTS AND LOCATIONS:
Overall Officials: Ya Mei Bai, M.D. Ph.D., Principal Investigator — Taipei Veterans General Hospital, Taiwan
Locations (1):
- Taipei Veterans General Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided